CLINICAL TRIAL: NCT05878002
Title: "Cognitive, Motor and Sleep Evaluation in Patients With Ischemic Stroke of Basal Ganglia After Thrombectomy"
Acronym: CMS - SBGT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5137
Record Dates: First submitted 2023-04-26; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-04

CONDITIONS: Post-stroke Disorders
MeSH Terms: interventions — Polysomnography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients affected by acute ischemic stroke treated with mechanical thrombectomy (Other)
  Interventions: Device: polysomnography

INTERVENTIONS:
Device: polysomnography — Sleep study through polysomnographic examination

SUMMARY:
The goal of this interventional study is to learn about the clinical outcomes of acute ischemic stroke treated with mechanical thrombectomy resulting in a selective ischemia of the basal ganglia. The main question it aims to answer is:

• defining the prevalence and clinical features of possible cognitive, motor and sleep disfuncions occuring after acute ischemic stroke treated with thrombectomy

Participants will be tested for cognitive, movement and sleep disorders in the acute phase and successively in the long term follow-up.

ELIGIBILITY:
Inclusion Criteria:

* participant's age ≥ 18 years
* acute ischemic stroke due to occlusion of proximal middle cerebral artery successfully treated with mechanical thrombectomy (mTICI ≥ 2B)
* signature of specific written informed consent

Exclusion Criteria:

* unstable clinical conditions
* personal history of cognitive decline before the acute ischemic stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2033-04-12 (Estimated); Study Completion 2034-04 (Estimated)

PRIMARY OUTCOMES:
Post-stroke cognitive dysfunction | Within 72 hours
  Assessment through the MoCA (Montreal Cognitive Assessment) score of cognitive dysfunction in patients with acute ischemic stroke treated with mechanical thrombectomy

CONTACTS AND LOCATIONS:
Locations (1):
- Flavia Torlizzi, Rome, Italy